CLINICAL TRIAL: NCT05055830
Title: Clinically Integrated Opportunistic PK/PD Trial in Critically Ill Children
Brief Title: Opportunistic PK/PD Trial in Critically Ill Children (OPTIC)
Acronym: OPTIC
Status: Recruiting | Type: Observational
Sponsor: Duke University (Other)
Collaborators: Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: Pro00108566
Record Dates: First submitted 2021-09-15; First posted 2021-09-24 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Cardiac Disease; Critically Ill; Children, Adult
MeSH Terms: conditions — Heart Diseases; Critical Illness | interventions — Methadone; Caffeine; Acetaminophen; Milrinone

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, effluent samples, tissue, and plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children (<21 years of age) who are prescribed drugs of interest: Children and young adults who are prescribed drugs of interest as part of their routine medical care and are admitted to the pediatric cardiac intensive care unit
  Interventions: Drug: The OPTIC study is collecting PK data on children prescribed understudied drugs of interest per standard of care.

INTERVENTIONS:
Drug: The OPTIC study is collecting PK data on children prescribed understudied drugs of interest per standard of care. — The goal of this study is to characterize the pharmacokinetics of understudied drugs for which specific dosing recommendations and safety data are lacking. The prescribing of drugs to children will not be part of this protocol. Taking advantage of procedures done as part of routine medical care (i.e. blood draws), this study will serve as a tool to better understand drug exposure in children receiving these drugs per standard of care.
  Other Names: Methadone; Caffeine; Acetaminophen; Milrinone

SUMMARY:
OPTIC is a prospective, open-label, non-randomized study of multiple medications administered to approximately 2000 children in the pediatric cardiac intensive care unit (PCICU) per routine clinical car by their treating provider. The purpose of this study is to characterize the PK of drugs routinely administered to children per standard of care using opportunistic and scavenged samples. The prescribing of drugs to children will not be part of this protocol.

After the child/adult (<21 years of age) is consented/enrolled, demographic and clinical data will be extracted from the EHR. Biospecimen information (including date and time of sample collection) will be collected.

Data analysis will be conducted on all participants with at least 2 evaluable samples. The protocol represents minimal risk to the children/adults who provide body fluid for this study, including potential loss of confidentiality (samples will be assigned a unique accession number) and risks associated with blood draws. Adverse Events (AEs)/Serious Adverse Events (SAEs) caused by the study specimen collections will be monitored and recorded in the Electronic Data Capture (EDC) system.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for enrollment, a potential participant must meet all the following criteria:

1. Participant is <21 years old on admission
2. Participant is admitted to the Pediatric Cardiac Intensive Care Unit
3. Parent/legal guardian/adult participant can understand the consent process and is willing to provide informed consent/assent
4. Participant is receiving one or more of the study drugs of interest at the time of enrollment

Exclusion Criteria:

1. Any condition which would make the participant, in the opinion of the investigator, unsuitable for the study

Ages: 0 Months to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children under 21 years of age
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2021-10-05 (Actual); Primary Completion 2027-10-30 (Estimated); Study Completion 2028-10-30 (Estimated)

PRIMARY OUTCOMES:
Clearance (CL) or apparent oral clearance (CL/F) as measured by PK sampling | Data will be collected up to 180 days from the time of consent
Half-life (t1/2) as measured by PK sampling | Data will be collected up to 180 days from the time of consent
Volume of distribution (V) or apparent oral volume of distribution (V/F) as measured by PK sampling | Data will be collected up to 180 days from the time of consent
AUC (area under the curve) as measured by PK sampling | Data will be collected up to 180 days from the time of consent

CONTACTS AND LOCATIONS:
Overall Officials: Christoph P Hornik, MD, PhD, MPH, Principal Investigator — Duke UMC
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Thompson EJ, Foote HP, Hill KD, Hornik CP. A point-of-care pharmacokinetic/pharmacodynamic trial in critically ill children: Study design and feasibility. Contemp Clin Trials Commun. 2023 Jul 7;35:101182. doi: 10.1016/j.conctc.2023.101182. eCollection 2023 Oct. PMID 37485397